CLINICAL TRIAL: NCT07125560
Title: The Effectiveness of Oral Health Education Module (MyBRUSH) in Improving Knowledge, Attitude, and Behaviour on Toothpaste Use and Toothbrushing Among 12-Year-Old Children in Tawau Division, Sabah: A Cluster Randomised Controlled Trial
Brief Title: Effectiveness MyBRUSH Module in Improving Knowledge, Attitude, and Behaviour on Toothpaste Use and Toothbrushing Among 12-Year-Old Children
Acronym: MyBRUSH module
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mohd Ritzuan Abdul Multalib, Dental Officer, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: USM/JEPeM/KK/24040379
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Oral Health; Knowledge; Attitude; Behavior; Dental Plaque
Keywords: Toothpastes; Toothbrushing; Children; Intervention effectiveness
MeSH Terms: conditions — Behavior; Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: MyBRUSH module
- Control group (Active Comparator)
  Interventions: Behavioral: BEGIN program

INTERVENTIONS:
Behavioral: MyBRUSH module — oral health education module that comprises of booklet for educational material, oral health talk, toothbrushing demonstration and return demonstration, and small group discussion
  Arms: Intervention group
Behavioral: BEGIN program — BEGIN program that comprise of toothbrushing demonstration and return demonstration
  Arms: Control group

SUMMARY:
The goal of this intervention study is to study the effectiveness of the oral health education module (MyBRUSH) in improving the knowledge, attitude, and behaviour on toothpaste use and toothbrushing among 12-year-old children. This study also aims to study the effectiveness of the MyBRUSH module in improving dental plaque among 12-year-old children. The main questions it aims to answer are:

1. Does the knowledge, attitude, and behaviour on toothpaste use and toothbrushing of 12-year-old children improve after receiving the MyBRUSH module?
2. Does the dental plaque score of 12-year-old children improve after receiving the MyBRUSH module?
3. Does the improvement in knowledge, attitude, and behaviour regarding toothpaste use and toothbrushing, as well as the dental plaque of 12-year-old children, be higher after receiving the MyBRUSH module compared to those who received the existing toothbrushing module?

Researchers will compare the MyBRUSH module to a BEGIN (existing toothbrushing module) to see if the MyBRUSH module is effective in improving the knowledge, attitude, and behaviour on toothpaste use and toothbrushing, as well as the dental plaque of 12-year-old children.

Participants will:

* A questionnaire will be used to assess knowledge, attitude, and behaviour regarding toothpaste use and toothbrushing. This assessment will be done at four time points (baseline, evaluation-1, evaluation-2, and evaluation-3), with a one-month interval between each time point.
* A group of participants will receive intervention based on MyBRUSH module and another group of participants will receive intervention based on BEGIN. Each intervention activity will be done after each evaluation assessment is completed.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian citizen
* Children born in 2013, who would be 12-year-old in 2025
* Children using toothpaste during toothbrushing

Exclusion Criteria:

- Children with special educational needs based on the Ministry of Education (MOE) Malaysia definition

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Knowledge, attitude, and behavior | Point measurement at baseline, evaluation-1, evaluation-2, and evaluation-3 with 1 month interval for each point measurement (total duration 4 months)
  Assessment of knowledge, attitude, and behavior on toothpaste use and toothbrushing using a questionnaire
Dental plaque score | Point measurement at baseline, evaluation-1, evaluation-2, and evaluation-3 with 1 month interval for each point measurement (total duration 4 months)
  Dental plaque score based on Silness and Löe plaque index

CONTACTS AND LOCATIONS:
Overall Officials: Mohd Ritzuan Abdul Multalib, Principal Investigator — Universiti Sains Malaysia
Locations (8):
- Malaysia (8):
  - SJKC Pai Sheng, Kunak, Sabah
  - SK Kampung Selamat, Kunak, Sabah
  - SK Mostyn, Kunak, Sabah
  - SK SKIM Kokos, Kunak, Sabah
  - SK Balung, Tawau, Sabah
  - SK Bombalai, Tawau, Sabah
  - SK Holy Trinity, Tawau, Sabah
  - SK Jambatan Putih, Tawau, Sabah

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR